CLINICAL TRIAL: NCT05360251
Title: Comparison of Efficacy and Safety of Pulsed Dye Laser and Intense Pulsed Light Configured With Different Wavelength Bands in the Treatment of Erythematotelangiectatic Rosacea
Brief Title: Pulsed Dye Laser and Intense Pulsed Light Configured With Different Wavelength Bands in Improving Erythematotelangiectatic Rosacea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-0177
Record Dates: First submitted 2022-04-30; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-03

CONDITIONS: Erythematotelangiectatic Rosacea
Keywords: Pulsed dye laser，intense pulse light
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Intervention Model Description: adult patients diagnosed with erythematotelangiectatic rosacea
Who Masked: Participant
Masking Description: patients are blinded to laser therapy received
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pulsed dye laser(PDL) (Experimental): The patients were randomly categorized into the following four groups based on the treatments they received: PDL, DPL, M22 590, M22 vascular filter
  Interventions: Device: PDL(595nm)
- IPL(Delicate Pulsed Light) (Experimental): The patients were randomly categorized into the following four groups based on the treatments they received: PDL, DPL, M22 590, M22 vascular filter
  Interventions: Device: IPL(DPL)
- IPL(M22 590) (Experimental): The patients were randomly categorized into the following four groups based on the treatments they received: PDL, DPL, M22 590, M22 vascular filter
  Interventions: Device: IPL(M22 590)
- IPL(M22 vascular filter) (Experimental): The patients were randomly categorized into the following four groups based on the treatments they received: PDL, DPL, M22 590, M22 vascular filter
  Interventions: Device: IPL(M22 vascular)

INTERVENTIONS:
Device: PDL(595nm) — One subject was treated with pulsed dye laser (Vbeam platinum, 595 nm, Candela Corporation): energy dosages of 9-11 J/cm2, pulse durations of 10/20 ms, and spot size of 7 mm.
  Arms: Pulsed dye laser(PDL)
Device: IPL(DPL) — One subject was treated with IPL(delicate Pulsed Light, Dye-VL, Alma Lasers Corporation): energy dosages of 8.4-10.6 J/cm2, pulse durations of 10/12 ms, and spot size of 10×30 mm.
  Arms: IPL(Delicate Pulsed Light)
Device: IPL(M22 590) — One subject was treated with IPL(M22 590, 590-1200nm, Lumenis Limited): energy dosages of 15-18 J/cm2, pulse durations of 3-4 ms, pulse delay of 30-40 ms, and spot size of 15×35 mm.
  Arms: IPL(M22 590)
Device: IPL(M22 vascular) — One subject was treated with IPL(M22 vascular, 530-650nm and 900-1200nm, Lumenis Limited): energy dosages of 9-17 J/cm2, pulse durations of 4-6 ms, pulse delay of 20-40 ms, and spot size of 15×35 mm.
  Arms: IPL(M22 vascular filter)

SUMMARY:
Pulsed dye laser(PDL) and intense pulsed light(IPL) has been widely used in improving rosacea. To compare the efficacy and safety of PDL and IPL configured with different wavelength bands(Delicate Pulsed Light, M22 590, M22 vascular filter) in the treatment of rosacea, we designed a prospective, randomized controlled trial. We hope to make a comparison between PDL and IPL,between broad-spectrum IPL and narrow-spectrum IPL, between single-band IPL and dual-band IPL, and also provide clinical basis for clinicians and patients to develop individualized treatment plans.

DETAILED DESCRIPTION:
Rosacea is a chronic skin condition characterized by erythema, inflammatory papules, pustules and telangiectasias, which typically occur on the face of middle-aged adults, especially fair skinned. The disease can lead to social stigmatization and may significantly reduce the quality of life of patients. For erythematous lesions and telangiectasia, intense pulsed light (IPL) therapy and lasers are popular treatmen option. Lasers and non-coherent intense pulse light sources (IPL) are based on the principle of selective photothermolysis. The target chromophore in vascular lesions is the oxyhemoglobin present in the red blood corpuscles (RBCs) which circulates in the blood vessels. Pulsed dye lasers (PDL) use a wavelength of 595 nm and is the gold standard of vascular lesion treatment. A common complication is post treatment purpura which appears immediately and can last for 7-14 days, which may be cosmetically unacceptable. The intense pulsed light (IPL) produces a non-coherent light beam with a spectrum of wavelengths from 500 to 1200 nm. Cut-off filters at 515, 550, 570, 590 nm are used for vascular lesions. To compare the efficacy and safety of PDL and IPL configured with different wavelength bands(Delicate Pulsed Light, M22 590, M22 vascular filter) in the treatment of rosacea, we designed a prospective, randomized controlled trial. We hope to make a comparison between PDL and IPL,between broad-spectrum IPL and narrow-spectrum IPL, between single-band IPL and dual-band IPL, and also provide clinical basis for clinicians and patients to develop individualized treatment plans.

ELIGIBILITY:
Inclusion Criteria:

age of at least 18 years; according to the rosacea diagnostic criteria established by the NRSEC in 2002, be diagnosed as erythematotelangiectatic rosacea; Rosacea clinical score is between 9 and 12; Fitzpatrick skin type III and IV;

Exclusion Criteria:

there was infection in the treatment site sunburn history within 1 month; received oral isotretinoin or laser treatment in the past 3 months received chemical peeling 1 month before the study pregnancy or breast-feeding. those who are receiving other treatment for rosacea, such as topical and oral drugs;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-27 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Rosacea clinical score | from baseline(T0) to 4weeks after the final treatment(T3)
  It includes objective symptom score(Flushing, Nontransient erythema, Telangiectasia) and subjective symptom score(Burning or stinging, Itching, Dry), with a 4-level score according to the standard grading system by NRS. Objective symptom is assessed by a dermatologist, and subjective symptom score is assessed by subjects themselves.
VISIA Red Area score | from baseline(T0) to 4weeks after the final treatment(T3)
  using VISIA image system to record red area absolute score

SECONDARY OUTCOMES:
Pain score | immediately after each laser treatment
  It is evaluated by subjects themselves with Visual analogue scale(VAS) , on a scale hypopigmentation were recorded.

OTHER OUTCOMES:
adverse effects | through study completion, an average of 0.5 year
  Adverse reactions such as pain, erythema and edema, hyperpigmentation and hypopigmentation were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Suiqing S Cai, doctor, Study Chair — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- The Second Affiliated Hospital of Zhejiang University of Medicine, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Since the individual participant data(IPD) is personal information, our participants are unwilling to share. But we welcome any questions through emails.

REFERENCES:
- [Derived] Ruan J, Zheng Y, Cai S. Efficacy and safety comparison between pulsed dye laser and intense pulsed light configured with different wavelength bands in treating erythematotelangiectatic rosacea. Lasers Med Sci. 2024 Jun 1;39(1):146. doi: 10.1007/s10103-024-04098-9. PMID 38822948